CLINICAL TRIAL: NCT02624622
Title: A Comparison Between Mothers and Community Health Workers on Use of Chlorhexidine for Umbilical Cord Care: A Randomized Noninferiority Trial
Brief Title: Chlorhexidine Cord Care for Newborn Infants in Kenya
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funds
Sponsor: University of New Mexico (Other)
Collaborators: University of Nairobi (Other)
Responsible Party: Principal Investigator, Angelo Tomedi, Principal Investigator, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UNM HRRC 14-356
Record Dates: First submitted 2015-12-03; First posted 2015-12-08 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Omphalitis
Keywords: omphalitis; neonate; developing countries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CHW applies chlorhexidine (Active Comparator): Intervention: Chlorhexidine gel 7.1% topical 3 gm applied to the umbilical cord stump in one application. The community health worker is given the chlorhexidine to apply to the umbilical cord stump within 24 hours of delivery of the newborn infant.
  Interventions: Procedure: Chlorhexidine application by CHW
- Mother applies chlorhexidine (Experimental): Intervention: Chlorhexidine gel 7.1% topical 3 gm applied to the umbilical cord stump in one application. Mother is given the chlorhexidine during the first prenatal care visit to apply to the umbilical cord stump within 24 hours of delivery of the newborn infant.
  Interventions: Procedure: Chlorhexidine application to cord by mother

INTERVENTIONS:
Procedure: Chlorhexidine application to cord by mother
  Arms: Mother applies chlorhexidine
Procedure: Chlorhexidine application by CHW
  Arms: CHW applies chlorhexidine

SUMMARY:
Studies in several countries with a high rate of death of infants during the first week of life have found a reduction in infection and mortality when chlorhexidine is applied to the umbilical cord stump by a health worker within 24 hours of birth. This study will evaluate if providing chlorhexidine to pregnant women during a prenatal care visit for application to the cord stump after birth will be as effective for preventing omphalitis (infection of the umbilical cord stump) as sending a community health worker into the home to apply the chlorhexidine.

DETAILED DESCRIPTION:
Neonatal mortality continues to be unacceptably high in Kenya and other Sub-Saharan African countries, with little improvement over the past several decades. Neonatal infections and sepsis are a leading cause of neonatal deaths. Three fourths of these deaths occur in the first week of life. Many deliveries in rural Kenya take place at home in unhygienic conditions and the umbilical cord is cut with unsterile instruments, increasing the risk of infection. Studies in several countries with a high neonatal mortality rate have found a reduction in infection and mortality when chlorhexidine is applied to the umbilical cord stump by a health worker within 24 hours of birth. This randomized noninferiority study in rural Kenya will compare the effectiveness of a newborn home visitation program that includes application of chlorhexidine to the umbilical cord by a visiting community health worker (CHW) to the provision of chlorhexidine to the mother during a prenatal care visit for cord application on the rate of omphalitis (infection of the umbilical cord stump) during the first week of life. Pregnant women will be randomly assigned in a 1:1 ration to be given or not be given chlorhexidine digluconate 7.1% gel during a prenatal care visit with instruction to apply the product as soon as possible after birth. The pregnant women who do not receive the chlorhexidine will be assigned a CHW with instruction to apply the product during a home visit within 24 hours of birth. The rate of omphalitis will be determined during home visits by the CHW on days three and seven after birth, and by a visiting research nurse on the seventh day. The time from birth to chlorhexidine application will also be recorded and compared in the two groups.

ELIGIBILITY:
Inclusion Criteria: All pregnant women who are 18 years of age or older (based on their stated date of birth) who attend the two selected health care facilities (Kisesini Dispensary and Katangi Health Center) for their prenatal care will be eligible to participate if they reside in one of the villages of the five sublocations of the target region (Kyua, Makusya, Katangi, Mekilingi, Syokisinga) and they plan to deliver within the target region -

Exclusion Criteria: Pregnant women who plan to deliver outside of the target area or plan to be away from the area during the newborn infant's first week of life will be excluded

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 576 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Number of infants age 0 to 7 days who develop omphalitis | 7 days after birth
  Omphalitis is defined as redness of the umbilical stump that extends to the skin of the abdomen with or without purulent exudate (pus).

SECONDARY OUTCOMES:
The average time in minutes from birth to chlorhexidine application (total time for all participants in the arm divided by total participants in the arm). | 7 days
  The duration in minutes from the recorded birth time until the recorded time that chlorhexidine is applied to the umbilical cord stump

CONTACTS AND LOCATIONS:
Overall Officials: ANGELO TOMEDI, MD, Principal Investigator — University of New Mexico
Locations (1):
- UNM, Albuquerque, New Mexico, United States